CLINICAL TRIAL: NCT04575012
Title: A Randomized Multicentre Trial to Compare Early With Deferred Invasive Strategy for Patients With Acute ST-segment Elevation Myocardial Infarction Presenting 24-48 Hours From Symptom Onset
Brief Title: Compare Early With Deferred Invasive Strategy for STEMI Presenting 24-48 Hours From Symptom Onset
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZS-STEMI 24-48
Record Dates: First submitted 2020-09-26; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: ST-segment Elevation Myocardial Infarction; Percutaneous Coronary Intervention; Invasive Strategy
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deferred invasive strategy (Experimental)
  Interventions: Procedure: Deferred invasive strategy
- Early invasive strategy (Other)
  Interventions: Procedure: Early invasive strategy

INTERVENTIONS:
Procedure: Deferred invasive strategy — PCI on 7 to 10 days after symptom onset
  Arms: Deferred invasive strategy
Procedure: Early invasive strategy — Primary PCI
  Arms: Early invasive strategy

SUMMARY:
The primary objective of the trial is to compare the efficacy of early with deferred invasive strategy for patients with ST-segment elevation myocardial infarction (STEMI) within 24-48h of symptom onset.

DETAILED DESCRIPTION:
At present, timely primary percutaneous coronary intervention (PCI) is the preferred strategy for STEMI patients within 24h of symptom onset. In stable STEMI patients presenting 12 to 48 hours from symptom onset, BRAVE-2 Trial (n = 365) showed improved myocardial salvage and 4-year survival in patients treated with primary PCI compared with conservative treatment alone. However, data is scarce about the reperfusion strategy focusing on STEMI patients within 24-48h of symptom onset.

To our knowledge, due to the long onset time and insufficient antiplatelet/anticoagulant treatment, infarct-related artery in STEMI patients beyond 24h of symptom onset frequently suffer from severer thrombus burden. In this situation, the risk of no-reflow in primary PCI is high. Meanwhile, myocardial coagulative necrosis would be fully developed during 24-72h from symptom onset, the risk of perioperative cardiac rupture may also rise. These bring some doubts about the benefits of early invasive strategy for STEMI patients within 24-48h of symptom onset. Further investigations are warranted to explore the best timing of invasive strategy for STEMI patients within 24-48h of symptom onset.

Given that no randomized clinical trial is designed especially for STEMI patients within 24-48h of symptom onset, and limited data is available to compare early with deferred invasive strategy for the subgroup of STEMI patients, investigators plan to perform a controlled, randomized trial to compare the efficacy of early with deferred invasive strategy for STEMI patients within 24-48h of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 or over and less than 75 years old;
2. ECG: ≥2 mm ST-segment elevation in 2 contiguous precordial leads or ≥1 mm ST-segment elevation in 2 contiguous extremity leads;
3. Patents with STEMI with symptom onset between 24 and 48 hours before randomization;
4. Signed informed consent form prior to trial participation.

Exclusion Criteria:

1. Patents with STEMI with symptom onset <24h or >48h or uncertain time onset;
2. Prior administration of thrombolytic therapy or attempted PCI before randomization;
3. Presence of indications for primary PCI, such as persistent chest pain, cardiogenic shock, life-threatening arrhythmias or cardiac arrest, severe acute heart failure, and mechanical complications;
4. Coagulopathy, active peptic ulcer, history of cerebral or subarachnoid hemorrhage, stroke within 6 months, other contraindications for antiplatelet or anticoagulant therapy;
5. Known intolerance to antiplatelet (e.g. aspirin, clopidogrel, ticagrelor) and anticoagulant therapy (e.g. heparin, bivalirudin);
6. Congenital heart disease or severe valvular disease;
7. eGFR <30 ml/min/1.73 m2;
8. History of malignant tumors;
9. Combined with other diseases and life expectancy ≤12 months;
10. Pregnancy;
11. Inclusion in another clinical trial;
12. Inability to provide informed consent or not available for follow-up judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
A composite of death from any cause, recurrent myocardial infarction, ischaemia-driven target vessel revascularization, or hospitalization due to NYHA class IV heart failure | 4 years

SECONDARY OUTCOMES:
No-reflow in infarct-related artery | Immediately after PCI
  The definition of no-reflow was Thrombolysis In Myocardial Infarction (TIMI) flow grade ≤ 2 on the final angiogram in a coronary angiographic analysis.
Major adverse cardiac events (defined as a composite of cardiac death, recurrent myocardial infarction, or ischaemia-driven target vessel revascularization) | 30 days
Stroke | 30 days
  The diagnosis of stroke required confirmation by computed tomography or magnetic resonance imaging of the head in the presence of a new onset focal or global neurological deficit lasting more than 24 hours.
Death from any cause | 4 years
Recurrent myocardial infarction | 4 years
Ischaemia-driven target vessel revascularization | 4 years
Hospitalization due to NYHA class IV heart failure | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, M.D., Principal Investigator — Shanghai Institute of Cardiovascular Diseases, Zhongshan Hospital, Fudan University

IPD SHARING:
Plan to Share IPD: No